CLINICAL TRIAL: NCT00174603
Title: Treatment of Major Depressive Disorder With Psychotic Features With Quetiapine Monotherapy; Quetiapine and Citalopram; or Haloperidol and Citalopram
Brief Title: Treatment of Depression With Quetiapine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: Rush University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRUSQUET305
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Major Depression With Psychotic Features
Keywords: depression; psychosis
MeSH Terms: conditions — Depression; Psychotic Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: quetiapine

SUMMARY:
The purpose of this study is to examine the mood stabilizing and antipsychotic properties of quetiapine in the treatment of depression by comparing subjects who were randomly assigned to either quetiapine monotherapy, quetiapine and citalopram; or haloperidol and citalopram. We hypothesize that quetiapine monotherapy would have similar effects to the combination of a first generation antipsychotic plus an antidepressant for the treatment of a major depressive episode with psychosis.

DETAILED DESCRIPTION:
Thus, current practice for treating psychotic depression is to combine an antidepressant with an antipsychotic. However, there are limitations to this approach. The rate of response is still lower than in other forms of major depression (Janicak et al., 2001). The rate of noncompliance is higher in this group; and the incidence of adverse effects related to the antipsychotic is increased (Janicak et al., 2001). As a result, studies have examined alternative treatments. The present study proposes to examine quetiapine's antipsychotic and mood stabilizing properties for the treatment of a major depressive disorder with psychotic features Subjects will be randomized to either quetipine monotherapy, quetiapine and citalopram; or haloperidol and citalopram.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 to 75 years.
* A Structured Clinical Interview for the DSM-IV (SCID) derived diagnosis of major depression with psychosis, single or recurrent episode (unipolar or bipolar).
* Subjects may have an anxiety disorder or an additional mood disorder such as dysthymia.
* Baseline 24-item Hamilton Depression Rating Scale (HDRS) score of greater than or equal to 21.
* A baseline Positive and Negative Syndrome Scale (PANSS) score of greater than or equal to 4 on at least one of the 4 psychosis items.
* Women of childbearing potential must agree to practice a medically accepted means of contraception.
* Length of current episode no longer than 3 months.

Exclusion Criteria:

* Pregnant or lactating women
* Women of child-bearing age who refuse a pregnancy test or who refuse to use a contraceptive technique when sexually active.
* Persons with other psychotic disorders; a mood disorder due to a general medical condition or substance-induced; substance dependence disorder in the last 6 months; substance abuse in the last 6 months or a dementing disorder are excluded.
* Persons with serious, unstable medical illnesses.
* Subjects who have been intolerant or nonresponsive to adequate trials of quetiapine, haloperidol and/or citalopram.
* Subjects who have received an injectable decanoate medication within 1 half life of the medication (i.e, 4 weeks for haloperidol or 2 weeks for fluphenazine).
* Subjects who have received fluoxetine within 4 weeks prior to randomization.
* Subjects who have received aripiprazole within 2 weeks prior to randomization.
* Subjects who have been treated with ECT within the last 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-08; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale
Young Mania Rating Scale
Barnes Akathisia Scale
Simpson Angus Scale
Clinical Global Impressions

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Janicak, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States